CLINICAL TRIAL: NCT04097821
Title: A Randomized, Open-label, Phase I/II Open Platform Study Evaluating Safety and Efficacy of Novel Ruxolitinib Combinations in Myelofibrosis Patients
Brief Title: Platform Study of Novel Ruxolitinib Combinations in Myelofibrosis Patients
Acronym: ADORE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC424H12201; 2019-000373-23 (EudraCT Number)
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Myelofibrosis
Keywords: myelofibrosis; ruxolitinib; INC424; siremadlin; HDM201; crizanlizumab; SEG101; sabatolimab; MBG453; rineterkib; LTT462; NIS793; platform study
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; siremadlin; crizanlizumab; sabatolimab; NIS-793

STUDY DESIGN:
Intervention Model Description: This open-label, multi-center, phase Ib/II platform study design consisted of 3 parts. Part 1 was a phase Ib dose escalation and safety run-in for the 5 novel agents in combination with ruxolitinib to assess safety, tolerability and to confirm recommended Phase II dose.
  Parts 2 and 3 were phase II selection and expansion respectively, to assess preliminary efficacy of the combination treatments from Part 1 that were evaluated as safe and tolerable.
  The number of combination treatment arms opening in Part 2 depended on the results of Part 1. In Part 2, interim analysis was planned to determine if combination treatment(s) could be expanded in Part 3.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1: Ruxolitinib + Siremadlin 20 mg (Experimental): Dose escalation of siremadlin added to existing stable dose of ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: Siremadlin
- Part 1: Ruxolitinib + Siremadlin 30 mg (Experimental): Dose escalation of siremadlin added to existing stable dose of ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: Siremadlin
- Part 1: Ruxolitinib + Siremadlin 40 mg (Experimental): Dose escalation of siremadlin added to existing stable dose of ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: Siremadlin
- Part 1: Ruxolitinib + Rineterkib 200 mg (Experimental): Dose escalation of rineterkib added to existing stable dose of ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: Rineterkib
- Part 1: Ruxolitinib + Crizanlizumab (Experimental): Safety run-in of crizanlizumab added to existing stable dose of ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: Crizanlizumab
- Part 1: Ruxolitinib + Sabatolimab (Experimental): Safety run-in of sabatolimab added to existing stable dose of ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: Sabatolimab
- Part 1: Ruxolitinib + NIS793 (Experimental): Safety run-in of NIS793 added to existing stable dose of ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: NIS793
- Part 2: Ruxolitinib (Active Comparator): Existing stable dose of ruxolitinib as control for Part 2
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablets for oral use
  Other Names: INC424, Jakavi
Drug: Siremadlin — 10 mg, 20 mg, or 40 mg capsules for oral use
  Other Names: HDM201
  Arms: Part 1: Ruxolitinib + Siremadlin 20 mg; Part 1: Ruxolitinib + Siremadlin 30 mg; Part 1: Ruxolitinib + Siremadlin 40 mg
Drug: Crizanlizumab — 100 mg/10 mL concentrate for infusion for intravenous use
  Other Names: SEG101
  Arms: Part 1: Ruxolitinib + Crizanlizumab
Drug: Sabatolimab — 100 mg/mL or 400 mg/4 mL concentrate for infusion for intravenous use
  Other Names: MBG453
  Arms: Part 1: Ruxolitinib + Sabatolimab
Drug: Rineterkib — 100 mg capsule for oral use
  Other Names: LTT462
  Arms: Part 1: Ruxolitinib + Rineterkib 200 mg
Drug: NIS793 — 700 mg/7 mL concentrate for infusion for intravenous use
  Arms: Part 1: Ruxolitinib + NIS793

SUMMARY:
The purpose of this study was to investigate the safety, pharmacokinetics and preliminary efficacy of combination treatment of ruxolitinib with 5 novel compounds: siremadlin, crizanlizumab, sabatolimab, rineterkib and NIS793 in myelofibrosis (MF) subjects.

DETAILED DESCRIPTION:
This open-label, multi-center, Phase Ib/II platform study design consisted of 3 parts. Part 1 was a Phase Ib dose escalation and safety run-in for the 5 novel agents in combination with ruxolitinib to assess safety, tolerability and to confirm a recommended Phase II dose. Dose escalation cohorts were treated with ruxoltinib + siremadlin or ruxolitinib + rineterkib. Safety run-in cohorts were treated with either ruxolitinb + sabatolimab, ruxolitinb + crizanlizumab or ruxolitinib + NIS7913.

Parts 2 and 3 were Phase II selection and expansion, respectively, to assess preliminary efficacy of the combination treatments from Part 1 that were evaluated as safe and tolerable. The number of combination treatment arms opening in Part 2 depended on the results of Part 1. In Part 2, an interim analysis was planned to determine if combination treatment(s) could be expanded in Part 3.

In June 2022, Novartis decided to permanently halt the study enrollment in all ongoing parts (Part 1 and Part 2), and Part 3 (expansion) was not initiated. With Protocol Amendment 8, an extension treatment phase of 12 cycles was added in Part 1 to allow access to the combination treatment for ongoing subjects deriving clinical benefit. In consideration of the enrollment halt, Parts 2 and 3 objectives were not pursued, and Part 1 objectives were updated accordingly.

ELIGIBILITY:
Core treatment phase Inclusion Criteria:

* Subjects have diagnosis of primary myelofibrosis (PMF) according to the 2016 World Health Organization (WHO) criteria, or diagnosis of post-essential thrombocythemia (ET) (PET-MF) or post-polycythemia vera (PV) myelofibrosis (PPV-MF) according to the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) 2007 criteria
* Palpable spleen of at least 5 cm from the left costal margin (LCM) to the point of greatest splenic protrusion or enlarged spleen volume of at least 450 cm3 per MRI or CT scan at baseline (a MRI/CT scan up to 8 weeks prior to first dose of study treatment can be accepted).
* Have been treated with ruxolitinib for at least 12 weeks prior to first dose of study treatment
* Are stable (no dose adjustments) on the prescribed ruxolitinib dose (between 5 and 25 mg twice a day (BID)) for ≥ 4 weeks prior to first dose of study treatment

Extension treatment phase inclusion criteria:

* Signed consent for the extension treatment phase
* ongoing in the core treatment phase
* demonstrates clinical benefit of treatment in core treatment phase per investigator's assessment.

Core treatment phase Exclusion Criteria:

* Not able to understand and to comply with study instructions and requirements.
* Received any investigational agent for the treatment of MF (except ruxolitinib) within 30 days of first dose of study treatment or within 5 half-lives of the study treatment, whichever is greater
* Peripheral blood blasts count of > 10%.
* has documented severe hypersensitivity reactions/immunogenicity (IG) to a prior biologic product or Received a monoclonal antibody (Ab) or immunoglobulin-based agent within 1 year of screening in NIS793, crizanlizumab or sabatolimab arms, or in rineterkib or siremadlin arms within <=4 weeks of screening or <=5 half-lives whichever is shorter
* Splenic irradiation within 6 months prior to the first dose of study drug
* Received blood platelet transfusion within 28 days prior to first dose of study treatment.

Extension treatment phase Exclusion Criteria:

* meets any of study treatment discontinuation criteria
* current evidence of treatment failure per investigator, following treatment in core treatment phase
* enrolled in another interventional study
* evidence of non-compliance to study procedures or withdrew consent in core treatment phase
* currently has unresolved toxicities for which study treatment has been interrupted in the core treatment phase
* local access to alternative myelofibrosis treatment including those currently under investigation in clinical trials as assessed suitable in the opinion of the investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Copenhagen, Denmark
- Germany (4):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Jena
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Florence, FI, Italy
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Spain (4):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- Switzerland (2):
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Kocaeli, Turkey (Türkiye)
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ross DM, Heidel FH, Perkins AC, Reiter A, Crodel C, Riley C, Gomez-Casares MT, Takacs I, Becker H, Lehmann T, Vinogradova O, Burbury K, Vannucchi AM, Gupta V, Wondergem M, Kiladjian JJ, Cleary G, Zhang A, Kota J, Prahallad A, Wroclawska M, Lu M, Harrison CN. ADORE: an open platform study of ruxolitinib in combination with other novel therapies in patients with myelofibrosis. Blood Adv. 2025 Aug 26;9(16):4195-4205. doi: 10.1182/bloodadvances.2025015860. PMID 40334082

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All inclusion and exclusion criteria were checked at screening.
Period: Overall Study
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793 | Part 2: Ruxolitinib
Started | 7 | 10 | 6 | 9 | 6 | 2 | 4 | 1
Completed | 6 | 8 | 2 | 6 | 4 | 0 | 3 | 0
Not Completed | 1 | 2 | 4 | 3 | 2 | 2 | 1 | 1
Not completed — Subject Decision | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1
Not completed — Death | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — New Therapy For Study Indication | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all subjects who received any study drug. Part 2 enrollment included 1 participant. Data are not reported for this participant in order to protect participant privacy and confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793 | Part 2: Ruxolitinib | Total
Number analyzed (Participants) | 7 | 10 | 6 | 9 | 6 | 2 | 4 | 0 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (6.5) | 62.3 (10.7) | 74.3 (9.9) | 67.3 (7.8) | 65.0 (8.1) | 62.5 (12.0) | 70.8 (7.3) |  | 67.4 (9.2)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 1 | 5 | 1 | 4 | 4 | 1 | 1 |  | 17
  >=65 | 6 | 5 | 5 | 5 | 2 | 1 | 3 |  | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 0 | 2 | 1 | 0 | 1 |  | 12
  Male | 5 | 4 | 6 | 7 | 5 | 2 | 3 |  | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 10 | 6 | 8 | 5 | 2 | 4 |  | 42
  Unknown | 0 | 0 | 0 | 1 | 1 | 0 | 0 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Dose Limiting Toxicities Within the First 2 Cycles in Part 1
Description: Incidence and severity of dose limiting toxicities within the first 2 cycles (6 or 8 weeks) in Part 1 of the study. DLTs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) criteria Version 5.0. Grade 0 was assigned for all non-missing values not graded as 1 or higher. Higher grade indicated more severity. Grade 5 was not used.
Time Frame: Baseline to the end of Cycle 2 (6 or 8 weeks)
Population: The dose-determining set included all subjects from the safety run-in and dose escalation part (Part 1) of the study who met the minimum exposure criterion and had sufficient safety evaluations or experienced a DLT between C1D1 and C3D1. Number analyzed is the number of participants with available data.
Measure: Number; unit: participants
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 6 | 7 | 5 | 9 | 5 | 2 | 0
participants
  Grade 3 | 0 | 0 | 1 | 1 | 0 | 0 |
  Grade 4 | 0 | 1 | 1 | 0 | 0 | 0 |

2. Primary Outcome: Response Rate at the End of Cycle 6 or Cycle 8 in Part 1
Description: Composite of anemia improvement (hemoglobin level) and no spleen volume progression and no symptom worsening in Part 2 and Part 3 of the study. For a subject to be considered a responder, all three components of the composite had to be fulfilled.
Time Frame: Baseline to the end of Cycle 6 or 8 (24 weeks)
Population: Enrollment was permanently halted; therefore, data were not collected for this outcome measure.
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Subjects Achieving an Improvement in Hemoglobin Level of ≥ 1.5 g/dL From Baseline in Part 1
Time Frame: Week 24, Week 48
Population: The full analysis set included all subjects who received any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 7 | 10 | 6 | 9 | 6 | 2 | 4
percentage of participants
  Week 24 | 0 | 0 | 0 | 11.1 | 16.7 | 0 | 0
  Week 48 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Subjects Achieving an Improvement in Hemoglobin Level of at Least >= 2.0 g/dL From Baseline in Part 1
Time Frame: Week 24, Week 48
Population: The full analysis set included all subjects who received any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 7 | 10 | 6 | 9 | 6 | 2 | 4
percentage of participants
  Week 24 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0
  Week 48 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0

5. Secondary Outcome: Change in Spleen Length From Baseline in Part 1
Description: Change in spleen length measured in centimeters by manual palpation.
Time Frame: Baseline, Week 24, Week 48
Population: The full analysis set included all subjects who received any study drug. Number analyzed is the number of participants with available data.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 6 | 8 | 4 | 4 | 4 | 0 | 0
centimeters
  Week 24 n=6,8,4,4,4,0,0 | -3.3 (2.6) | -5.5 (3.9) | -6.3 (4.6) | -1.8 (3.9) | -1.5 (1.9) |  |
  Week 48 n=2,1,2,1,1,0,0: number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 0 | 0
  Week 48 n=2,1,2,1,1,0,0 | -5.0 (0.0) | -9.0 (NA) — Standard deviation was not calculable due to the single data point. | -6.0 (7.1) | -8.0 (NA) — Standard deviation was not calculable due to the single data point. | -5.0 (NA) — Standard deviation was not calculable due to the single data point. |  |

6. Secondary Outcome: Percentage of Subjects With >=35% Reduction in Spleen Volume From Baseline in Part 1
Description: Change in spleen volume measured by magnetic resonance imaging (MRI) or computed tomography (CT) from baseline.
Time Frame: Week 24, Week 48
Population: The full analysis set included all subjects who received any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 7 | 10 | 6 | 9 | 6 | 2 | 4
percentage of participants
  Week 24 | 14.3 | 60.0 | 0 | 0 | 0 | 0 | 0
  Week 48 | 14.3 | 10.0 | 16.7 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Subjects With >=25% Reduction in Spleen Volume From Baseline in Part 1
Description: Change in spleen volume measured by magnetic resonance imaging (MRI) or computed tomography (CT) from baseline.
Time Frame: Week 24, Week 48
Population: The full analysis set included all subjects who received any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 7 | 10 | 6 | 9 | 6 | 2 | 4
percentage of participants
  Week 24 | 28.6 | 60.0 | 0 | 11.1 | 0 | 0 | 0
  Week 48 | 28.6 | 10.0 | 16.7 | 11.1 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Subjects in Part 1 With >=50% Reduction From Baseline in Myelofibrosis Symptom Assessment Form, Version 4.0 (MFSAF v4.0)
Description: The MFSAF v4.0 questionnaire focuses on the 7 core symptoms of MF: fatigue, night sweats, pruritus, abdominal discomfort, pain under the ribs on the left side, early satiety and bone pain. Subjects record symptom severity at it worst for each of the 7 symptoms on an 11-point numeric rating scale, from 0 (absent) to 10 (worst imaginable). The Total Symptom Score (TSS) is the sum of all the scores for all 7 symptoms.
Time Frame: Week 12, Week 24, Week 48
Population: The full analysis set included all subjects who received any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 7 | 10 | 6 | 9 | 6 | 2 | 4
percentage of participants
  Week 12 | 42.9 | 30.0 | 16.7 | 11.1 | 16.7 | 0 | 0
  Week 24 | 14.3 | 20.0 | 33.3 | 11.1 | 16.7 | 0 | 0
  Week 48 | 14.3 | 10.0 | 16.7 | 0 | 0 | 0 | 0

9. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) for Siremadlin, Rineterkib, Crizanlizumab, Sabatolimab, and NIS793 in Part 1
Time Frame: Days 1 and 5 of Cycles 1 and 2 for siremadlin and Cycles 1 and 3 for crizanlizumab, sabatolimab, and NIS793; Days 1 and 15 of Cycle 1 for rineterkib
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Part 1: Ruxolitinib + Siremadlin 20 mg (AUClast for Siremadlin); Part 1: Ruxolitinib + Siremadlin 30 mg (AUClast for Siremadlin); Part 1: Ruxolitinib + Siremadlin 40 mg (AUClast for Siremadlin): Dose escalation of siremadlin added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Rineterkib 200 mg (AUClast for Rineterkib): Dose escalation of rineterkib added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Crizanlizumab (AUClast for Crizanlizumab): Safety run-in of crizanlizumab added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Sabatolimab (AUClast for Sabatolimab): Safety run-in of sabatolimab added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + NIS793 (AUClast for NIS793): Safety run-in of NIS793 added to existing stable dose of ruxolitinib
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg (AUClast for Siremadlin) | Part 1: Ruxolitinib + Siremadlin 30 mg (AUClast for Siremadlin) | Part 1: Ruxolitinib + Siremadlin 40 mg (AUClast for Siremadlin) | Part 1: Ruxolitinib + Rineterkib 200 mg (AUClast for Rineterkib) | Part 1: Ruxolitinib + Crizanlizumab (AUClast for Crizanlizumab) | Part 1: Ruxolitinib + Sabatolimab (AUClast for Sabatolimab) | Part 1: Ruxolitinib + NIS793 (AUClast for NIS793)
Number analyzed (Participants) | 6 | 9 | 5 | 9 | 5 | 2 | 4
ng*hr/mL
  Cycle 1 Day 1 n=6,9,5,9,5,2,4 | 1520 (619) | 2560 (1530) | 3780 (1840) | 6000 (5120) | 14100000 (4990000) | 34900 (7860) | 103000000 (18700000)
  Cycle 1 Day 5 n=6,7,5,0,0,0,0: number analyzed (Participants) | 6 | 7 | 5 | 0 | 0 | 0 | 0
  Cycle 1 Day 5 n=6,7,5,0,0,0,0 | 2230 (1110) | 3340 (2120) | 4390 (2270) |  |  |  |
  Cycle 2 Day 1 n=5,6,3,0,0,0,0: number analyzed (Participants) | 5 | 6 | 3 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 n=5,6,3,0,0,0,0 | 1720 (1020) | 2400 (1150) | 2870 (326) |  |  |  |
  Cycle 2 Day 5 n=3,5,3,0,0,0,0: number analyzed (Participants) | 3 | 5 | 3 | 0 | 0 | 0 | 0
  Cycle 2 Day 5 n=3,5,3,0,0,0,0 | 1590 (577) | 2860 (1680) | 3030 (786) |  |  |  |
  Cycle 1 Day 15 n=0,0,0,9,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 9 | 0 | 0 | 0
  Cycle 1 Day 15 n=0,0,0,9,0,0,0 |  |  |  | 15800 (11000) |  |  |
  Cycle 3 Day 1 n=0,0,0,0,5,2,3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 2 | 3
  Cycle 3 Day 1 n=0,0,0,0,5,2,3 |  |  |  |  | 20900000 (13000000) | 43500 (9110) | 166000000 (63600000)

10. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) for Ruxolitinib in Part 1
Time Frame: Days 1 and 5 of Cycles 1 and 2; Day 15 of Cycle 1
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 3 | 4 | 2 | 3 | 2 | 2 | 2
ng*hr/mL
  Ruxolitinib 5 mg Cycle 1 Day 1 n=0,0,2,1,0,0,0: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 1 n=0,0,2,1,0,0,0 |  |  | 344 (225) | 199 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 1 n=3,4,1,2,1,2,1: number analyzed (Participants) | 3 | 4 | 1 | 2 | 1 | 2 | 1
  Ruxolitinib 10 mg Cycle 1 Day 1 n=3,4,1,2,1,2,1 | 546 (412) | 673 (290) | 498 (NA) — Standard deviation was not calculable due to the single data point. | 633 (393) | 440 (NA) — Standard deviation was not calculable due to the single data point. | 336 (30.6) | 452 (NA) — Standard deviation was not calculable due to the single data point.
  Ruxolitinib 15 mg Cycle 1 Day 1 n=1,0,2,1,2,0,2: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 0 | 2
  Ruxolitinib 15 mg Cycle 1 Day 1 n=1,0,2,1,2,0,2 | 1090 (NA) — Standard deviation was not calculable due to the single data point. |  | 481 (243) | 729 (NA) — Standard deviation was not calculable due to the single data point. | 662 (420) |  | 1220 (637)
  Ruxolitinib 20 mg Cycle 1 Day 1 n=3,2,1,3,1,0,0: number analyzed (Participants) | 3 | 2 | 1 | 3 | 1 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 1 n=3,2,1,3,1,0,0 | 991 (183) | 616 (107) | 623 (NA) — Standard deviation was not calculable due to the single data point. | 913 (451) | 887 (NA) — Standard deviation was not calculable due to the single data point. |  |
  Ruxolitinib 25 mg Cycle 1 Day 1 n=0,0,0,1,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Ruxolitinib 25 mg Cycle 1 Day 1 n=0,0,0,1,0,0,1 |  |  |  | 188 (NA) — Standard deviation was not calculable due to the single data point. |  |  | 859 (NA) — Standard deviation was not calculable due to the single data point.
  Ruxolitinib 5 mg Cycle 1 Day 5 n=0,0,2,0,0,0,0: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 5 n=0,0,2,0,0,0,0 |  |  | 245 (173) |  |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 5 n=3,3,1,0,0,0,0,: number analyzed (Participants) | 3 | 3 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 1 Day 5 n=3,3,1,0,0,0,0, | 465 (228) | 550 (307) | 441 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 15 mg Cycle 1 Day 5 n=1,1,2,0,0,0,0: number analyzed (Participants) | 1 | 1 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 1 Day 5 n=1,1,2,0,0,0,0 | 849 (NA) — Standard deviation was not calculable due to the single data point. | 901 (NA) — Standard deviation was not calculable due to the single data point. | 454 (212) |  |  |  |
  Ruxolitinib 20 mg Cycle 1 Day 5 n=2,4,1,0,0,0,0: number analyzed (Participants) | 2 | 4 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 5 n=2,4,1,0,0,0,0 | 872 (218) | 652 (218) | 482 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 5 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 289 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 15 n=0,0,0,2,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 1 Day 15 n=0,0,0,2,0,0,0 |  |  |  | 592 (403) |  |  |
  Ruxolitinib 15 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0,: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0, |  |  |  | 518 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 20 mg Cycle 1 Day 15 n=0,0,0,3,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 15 n=0,0,0,3,0,0,0 |  |  |  | 957 (479) |  |  |
  Ruxolitinib 25 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 25 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 718 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 5 mg Cycle 2 Day 1 n=0,0,1,0,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 2 Day 1 n=0,0,1,0,0,0,0 |  |  | 172 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 10 mg Cycle 2 Day 1 n=2,2,1,0,0,0,0: number analyzed (Participants) | 2 | 2 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 2 Day 1 n=2,2,1,0,0,0,0 | 354 (101) | 507 (225) | 553 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 15 mg Cycle 2 Day 1 n=1,2,2,0,0,0,0: number analyzed (Participants) | 1 | 2 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 2 Day 1 n=1,2,2,0,0,0,0 | 1040 (NA) — Standard deviation was not calculable due to the single data point. | 1190 (214) | 334 (98.7) |  |  |  |
  Ruxolitinib 20 mg Cycle 2 Day 1 n=3,3,1,0,0,0,0: number analyzed (Participants) | 3 | 3 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 2 Day 1 n=3,3,1,0,0,0,0 | 823 (206) | 727 (200) | 521 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |

11. Secondary Outcome: Maximum (Peak) Observed Plasma Drug Concentration (Cmax) for Siremadlin, Rineterkib, Crizanlizumab, Sabatolimab, and NIS793 in Part 1
Time Frame: as for outcome 9
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1: Ruxolitinib + Siremadlin 20 mg (Cmax for Siremadlin); Part 1: Ruxolitinib + Siremadlin 30 mg (Cmax for Siremadlin); Part 1: Ruxolitinib + Siremadlin 40 mg (Cmax for Siremadlin): Dose escalation of siremadlin added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Rineterkib 200 mg (Cmax for Rineterkib): Dose escalation of rineterkib added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Crizanlizumab (Cmax for Crizanlizumab): Safety run-in of crizanlizumab added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Sabatolimab (Cmax for Sabatolimab): Safety run-in of sabatolimab added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + NIS793 (Cmax for NIS793): Safety run-in of NIS793 added to existing stable dose of ruxolitinib
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg (Cmax for Siremadlin) | Part 1: Ruxolitinib + Siremadlin 30 mg (Cmax for Siremadlin) | Part 1: Ruxolitinib + Siremadlin 40 mg (Cmax for Siremadlin) | Part 1: Ruxolitinib + Rineterkib 200 mg (Cmax for Rineterkib) | Part 1: Ruxolitinib + Crizanlizumab (Cmax for Crizanlizumab) | Part 1: Ruxolitinib + Sabatolimab (Cmax for Sabatolimab) | Part 1: Ruxolitinib + NIS793 (Cmax for NIS793)
Number analyzed (Participants) | 6 | 9 | 5 | 9 | 5 | 2 | 4
ng/mL
  Cycle 1 Day 1 n=6,9,5,9,5,2,4 | 118 (32.8) | 207 (122) | 290 (56.1) | 469 (358) | 114000 (36400) | 131 (17.7) | 439000 (56100)
  Cycle 1 Day 5 n=6,7,5,0,0,0,0: number analyzed (Participants) | 6 | 7 | 5 | 0 | 0 | 0 | 0
  Cycle 1 Day 5 n=6,7,5,0,0,0,0 | 161 (78.0) | 284 (138) | 336 (109) |  |  |  |
  Cycle 2 Day 1 n=5,6,3,0,0,0,0: number analyzed (Participants) | 5 | 6 | 3 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 n=5,6,3,0,0,0,0 | 131 (57.9) | 142 (102) | 268 (15.0) |  |  |  |
  Cycle 2 Day 5 n=3,5,3,0,0,0,0: number analyzed (Participants) | 3 | 5 | 3 | 0 | 0 | 0 | 0
  Cycle 2 Day 5 n=3,5,3,0,0,0,0 | 103 (34.1) | 193 (95.0) | 228 (58.3) |  |  |  |
  Cycle 1 Day 15 n=0,0,0,9,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 9 | 0 | 0 | 0
  Cycle 1 Day 15 n=0,0,0,9,0,0,0 |  |  |  | 987 (621) |  |  |
  Cycle 3 Day 1 n=0,0,0,0,5,2,3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 2 | 3
  Cycle 3 Day 1 n=0,0,0,0,5,2,3 |  |  |  |  | 114000 (56600) | 150 (33.2) | 743000 (314000)

12. Secondary Outcome: Maximum (Peak) Observed Plasma Drug Concentration (Cmax) for Ruxolitinib in Part 1
Time Frame: Days 1 and 5 of Cycles 1 and 2; Day 15 of Cycle 1
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 3 | 4 | 2 | 3 | 2 | 2 | 2
ng/mL
  Ruxolitinib 5 mg Cycle 1 Day 1 n=0,0,2,1,0,0,0: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 1 n=0,0,2,1,0,0,0 |  |  | 93.3 (26.5) | 67.4 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 1 n=3,4,1,2,1,2,1: number analyzed (Participants) | 3 | 4 | 1 | 2 | 1 | 2 | 1
  Ruxolitinib 10 mg Cycle 1 Day 1 n=3,4,1,2,1,2,1 | 184 (159) | 209 (20.8) | 108 (NA) — Standard deviation was not calculable due to the single data point. | 195 (41.0) | 191 (NA) — Standard deviation was not calculable due to the single data point. | 118 (33.0) | 132 (NA) — Standard deviation was not calculable due to the single data point.
  Ruxolitinib 15 mg Cycle 1 Day 1 n=1,0,2,1,2,0,2: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 0 | 2
  Ruxolitinib 15 mg Cycle 1 Day 1 n=1,0,2,1,2,0,2 | 334 (NA) — Standard deviation was not calculable due to the single data point. |  | 119 (76.2) | 193 (NA) — Standard deviation was not calculable due to the single data point. | 185 (120) |  | 254 (73.5)
  Ruxolitinib 20 mg Cycle 1 Day 1 n=3,2,1,3,1,0,0: number analyzed (Participants) | 3 | 2 | 1 | 3 | 1 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 1 n=3,2,1,3,1,0,0 | 310 (131) | 184 (14.8) | 232 (NA) — Standard deviation was not calculable due to the single data point. | 332 (33.5) | 221 (NA) — Standard deviation was not calculable due to the single data point. |  |
  Ruxolitinib 25 mg Cycle 1 Day 1 n=0,0,0,1,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Ruxolitinib 25 mg Cycle 1 Day 1 n=0,0,0,1,0,0,1 |  |  |  | 46.0 (NA) — Standard deviation was not calculable due to the single data point. |  |  | 224 (NA) — Standard deviation was not calculable due to the single data point.
  Ruxolitinib 5 mg Cycle 1 Day 5 n=0,0,2,0,0,0,0: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 5 n=0,0,2,0,0,0,0 |  |  | 74.8 (13.5) |  |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 5 n=3,3,1,0,0,0,0: number analyzed (Participants) | 3 | 3 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 1 Day 5 n=3,3,1,0,0,0,0 | 152 (55.3) | 149 (67.6) | 107 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 15 mg Cycle 1 Day 5 n=1,1,2,0,0,0,0: number analyzed (Participants) | 1 | 1 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 1 Day 5 n=1,1,2,0,0,0,0 | 252 (NA) — Standard deviation was not calculable due to the single data point. | 264 (NA) — Standard deviation was not calculable due to the single data point. | 172 (96.9) |  |  |  |
  Ruxolitinib 20 mg Cycle 1 Day 5 n=2,4,1,0,0,0,0: number analyzed (Participants) | 2 | 4 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 5 n=2,4,1,0,0,0,0 | 211 (48.8) | 232 (104) | 180 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 5 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 95.4 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 15 n=0,0,0,2,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 1 Day 15 n=0,0,0,2,0,0,0 |  |  |  | 158 (68.6) |  |  |
  Ruxolitinib 15 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 126 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 20 mg Cycle 1 Day 15 n=0,0,0,3,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 15 n=0,0,0,3,0,0,0 |  |  |  | 369 (83.7) |  |  |
  Ruxolitinib 25 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 25 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 323 (NA) — Standard deviation was not calculable due to the single data point. |  |  |
  Ruxolitinib 5 mg Cycle 2 Day 1 n=0,0,1,0,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 2 Day 1 n=0,0,1,0,0,0,0 |  |  | 82.1 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 10 mg Cycle 2 Day 1 n=2,2,1,0,0,0,0: number analyzed (Participants) | 2 | 2 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 2 Day 1 n=2,2,1,0,0,0,0 | 119 (66.7) | 165 (29.7) | 90.5 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |
  Ruxolitinib 15 mg Cycle 2 Day 1 n=1,2,2,0,0,0,0: number analyzed (Participants) | 1 | 2 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 2 Day 1 n=1,2,2,0,0,0,0 | 260 (NA) — Standard deviation was not calculable due to the single data point. | 337 (70.7) | 100 (68.9) |  |  |  |
  Ruxolitinib 20 mg Cycle 2 Day 1 n=3,3,1,0,0,0,0: number analyzed (Participants) | 3 | 3 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 2 Day 1 n=3,3,1,0,0,0,0 | 257 (71.0) | 176 (66.0) | 241 (NA) — Standard deviation was not calculable due to the single data point. |  |  |  |

13. Secondary Outcome: Time to Reach Maximum (Peak) Plasma, Blood, Serum or Other Body Fluid Drug Concentration After Single Dose Administration (Tmax) for Siremadlin, Rineterkib, Crizanlizumab, Sabatolimab, and NIS793 in Part 1
Time Frame: as for outcome 9
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Median (Full Range); unit: hours
Groups:
- Part 1: Ruxolitinib + Siremadlin 20 mg (Tmax for Siremadlin); Part 1: Ruxolitinib + Siremadlin 30 mg (Tmax for Siremadlin); Part 1: Ruxolitinib + Siremadlin 40 mg (Tmax for Siremadlin): Dose escalation of siremadlin added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Rineterkib 200 mg (Tmax for Rineterkib): Dose escalation of rineterkib added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Crizanlizumab (Tmax for Crizanlizumab): Safety run-in of crizanlizumab added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + Sabatolimab (Tmax for Sabatolimab): Safety run-in of sabatolimab added to existing stable dose of ruxolitinib
- Part 1: Ruxolitinib + NIS793 (Tmax for NIS793): Safety run-in of NIS793 added to existing stable dose of ruxolitinib
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg (Tmax for Siremadlin) | Part 1: Ruxolitinib + Siremadlin 30 mg (Tmax for Siremadlin) | Part 1: Ruxolitinib + Siremadlin 40 mg (Tmax for Siremadlin) | Part 1: Ruxolitinib + Rineterkib 200 mg (Tmax for Rineterkib) | Part 1: Ruxolitinib + Crizanlizumab (Tmax for Crizanlizumab) | Part 1: Ruxolitinib + Sabatolimab (Tmax for Sabatolimab) | Part 1: Ruxolitinib + NIS793 (Tmax for NIS793)
Number analyzed (Participants) | 6 | 9 | 5 | 9 | 5 | 2 | 4
hours
  Cycle 1 Day 1 n=6,9,5,9,5,2,4 | 2.52 [1.83 to 23.5] | 3.00 [1.92 to 7.45] | 3.93 [2.00 to 8.00] | 3.92 [1.98 to 24.0] | 1.82 [1.50 to 2.27] | 1.84 [1.67 to 2.00] | 2.00 [1.95 to 2.98]
  Cycle 1 Day 5 n=6,7,5,0,0,0,0: number analyzed (Participants) | 6 | 7 | 5 | 0 | 0 | 0 | 0
  Cycle 1 Day 5 n=6,7,5,0,0,0,0 | 3.44 [1.83 to 4.07] | 2.90 [2.00 to 3.97] | 2.87 [1.88 to 3.03] |  |  |  |
  Cycle 2 Day 1 n=5,6,3,0,0,0,0: number analyzed (Participants) | 5 | 6 | 3 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 n=5,6,3,0,0,0,0 | 1.95 [0.980 to 4.10] | 3.92 [2.83 to 23.9] | 2.88 [2.08 to 7.07] |  |  |  |
  Cycle 2 Day 5 n=3,5,3,0,0,0,0: number analyzed (Participants) | 3 | 5 | 3 | 0 | 0 | 0 | 0
  Cycle 2 Day 5 n=3,5,3,0,0,0,0 | 3.00 [2.95 to 3.17] | 2.93 [2.75 to 3.17] | 3.02 [2.92 to 3.08] |  |  |  |
  Cycle 1 Day 15 n=0,0,0,9,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 9 | 0 | 0 | 0
  Cycle 1 Day 15 n=0,0,0,9,0,0,0 |  |  |  | 2.50 [0.500 to 4.00] |  |  |
  Cycle 3 Day 1 n=0,0,0,0,5,2,3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 2 | 3
  Cycle 3 Day 1 n=0,0,0,0,5,2,3 |  |  |  |  | 1.65 [0.750 to 2.13] | 2.01 [1.85 to 2.17] | 1.97 [1.92 to 2.33]

14. Secondary Outcome: Time to Reach Maximum (Peak) Plasma, Blood, Serum or Other Body Fluid Drug Concentration After Single Dose Administration (Tmax) for Ruxolitinib in Part 1
Time Frame: Days 1 and 5 of Cycles 1 and 2; Day 15 of Cycle 1
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 3 | 4 | 2 | 3 | 2 | 2 | 2
hours
  Ruxolitinib 5 mg Cycle 1 Day 1 n=0,0,2,1,0,0,0: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 1 n=0,0,2,1,0,0,0 |  |  | 0.960 [0.920 to 1.00] | 0.500 [0.500 to 0.500] |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 1 n=3,4,1,2,1,2,1: number analyzed (Participants) | 3 | 4 | 1 | 2 | 1 | 2 | 1
  Ruxolitinib 10 mg Cycle 1 Day 1 n=3,4,1,2,1,2,1 | 0.550 [0.330 to 6.18] | 0.775 [0.500 to 1.08] | 0.500 [0.500 to 0.500] | 0.485 [0.470 to 0.500] | 0.580 [0.580 to 0.580] | 0.460 [0.00 to 0.920] | 1.67 [1.67 to 1.67]
  Ruxolitinib 15 mg Cycle 1 Day 1 n=1,0,2,1,2,0,2: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 0 | 2
  Ruxolitinib 15 mg Cycle 1 Day 1 n=1,0,2,1,2,0,2 | 0.650 [0.650 to 0.650] |  | 1.96 [1.92 to 2.00] | 0.420 [0.420 to 0.420] | 1.80 [1.75 to 1.85] |  | 2.42 [1.08 to 3.75]
  Ruxolitinib 20 mg Cycle 1 Day 1 n=3,2,1,3,1,0,0: number analyzed (Participants) | 3 | 2 | 1 | 3 | 1 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 1 n=3,2,1,3,1,0,0 | 0.530 [0.500 to 1.00] | 1.54 [1.08 to 2.00] | 1.00 [1.00 to 1.00] | 0.450 [0.420 to 1.03] | 1.17 [1.17 to 1.17] |  |
  Ruxolitinib 25 mg Cycle 1 Day 1 n=0,0,0,1,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Ruxolitinib 25 mg Cycle 1 Day 1 n=0,0,0,1,0,0,1 |  |  |  | 0.00 [0.00 to 0.00] |  |  | 2.00 [2.00 to 2.00]
  Ruxolitinib 5 mg Cycle 1 Day 5 n=0,0,2,0,0,0,0: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 5 n=0,0,2,0,0,0,0 |  |  | 0.960 [0.920 to 1.00] |  |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 5 n=3,3,1,0,0,0,0: number analyzed (Participants) | 3 | 3 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 1 Day 5 n=3,3,1,0,0,0,0 | 1.00 [0.830 to 2.02] | 0.980 [0.920 to 2.03] | 1.00 [1.00 to 1.00] |  |  |  |
  Ruxolitinib 15 mg Cycle 1 Day 5 n=1,1,2,0,0,0,0: number analyzed (Participants) | 1 | 1 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 1 Day 5 n=1,1,2,0,0,0,0 | 0.970 [0.970 to 0.970] | 0.830 [0.830 to 0.830] | 0.955 [0.830 to 1.08] |  |  |  |
  Ruxolitinib 20 mg Cycle 1 Day 5 n=2,4,1,0,0,0,0: number analyzed (Participants) | 2 | 4 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 5 n=2,4,1,0,0,0,0 | 0.925 [0.850 to 1.00] | 1.00 [0.920 to 1.08] | 0.830 [0.830 to 0.830] |  |  |  |
  Ruxolitinib 5 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 0.500 [0.500 to 0.500] |  |  |
  Ruxolitinib 10 mg Cycle 1 Day 15 n=0,0,0,2,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 1 Day 15 n=0,0,0,2,0,0,0 |  |  |  | 1.98 [1.95 to 2.00] |  |  |
  Ruxolitinib 15 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 0.500 [0.500 to 0.500] |  |  |
  Ruxolitinib 20 mg Cycle 1 Day 15 n=0,0,0,3,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 1 Day 15 n=0,0,0,3,0,0,0 |  |  |  | 0.650 [0.500 to 1.00] |  |  |
  Ruxolitinib 25 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ruxolitinib 25 mg Cycle 1 Day 15 n=0,0,0,1,0,0,0 |  |  |  | 0.500 [0.500 to 0.500] |  |  |
  Ruxolitinib 5 mg Cycle 2 Day 1 n=0,0,1,0,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 5 mg Cycle 2 Day 1 n=0,0,1,0,0,0,0 |  |  | 0.900 [0.900 to 0.900] |  |  |  |
  Ruxolitinib 10 mg Cycle 2 Day 1 n=2,2,1,0,0,0,0: number analyzed (Participants) | 2 | 2 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 10 mg Cycle 2 Day 1 n=2,2,1,0,0,0,0 | 0.895 [0.870 to 0.920] | 1.00 [0.920 to 1.08] | 2.00 [2.00 to 2.00] |  |  |  |
  Ruxolitinib 15 mg Cycle 2 Day 1 n=1,2,2,0,0,0,0: number analyzed (Participants) | 1 | 2 | 2 | 0 | 0 | 0 | 0
  Ruxolitinib 15 mg Cycle 2 Day 1 n=1,2,2,0,0,0,0 | 1.05 [1.05 to 1.05] | 1.46 [1.00 to 1.92] | 4.00 [0.920 to 7.07] |  |  |  |
  Ruxolitinib 20 mg Cycle 2 Day 1 n=3,3,1,0,0,0,0: number analyzed (Participants) | 3 | 3 | 1 | 0 | 0 | 0 | 0
  Ruxolitinib 20 mg Cycle 2 Day 1 n=3,3,1,0,0,0,0 | 0.980 [0.880 to 1.02] | 1.02 [1.00 to 4.00] | 0.930 [0.930 to 0.930] |  |  |  |

15. Secondary Outcome: Concentration Versus Time Profile for Siremadlin in Part 1
Time Frame: Day 1 of Cycles 1 and 2; Day 6 of Cycle 1; Days 2 and 5 of Cycles 1, 2, 3, 4, 5, and 6. Each cycle was 28 days.
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg
Number analyzed (Participants) | 7 | 10 | 5
ng/mL
  Cycle 1 Day 1, 0 hr (pre-dose) n=6,7,5: number analyzed (Participants) | 6 | 7 | 5
  Cycle 1 Day 1, 0 hr (pre-dose) n=6,7,5 | 0 (0) | 0 (0) | 0 (0)
  Cycle 1 Day 1, 0.5 hr n=6,8,5: number analyzed (Participants) | 6 | 8 | 5
  Cycle 1 Day 1, 0.5 hr n=6,8,5 | 7.46 (6.23) | 4.76 (8.02) | 12.8 (21.0)
  Cycle 1 Day 1, 1 hr n=6,9,5: number analyzed (Participants) | 6 | 9 | 5
  Cycle 1 Day 1, 1 hr n=6,9,5 | 52.7 (27.0) | 38.8 (40.9) | 87.0 (73.6)
  Cycle 1 Day 1, 2 hr n=6,9,5: number analyzed (Participants) | 6 | 9 | 5
  Cycle 1 Day 1, 2 hr n=6,9,5 | 104 (53.3) | 146 (95.1) | 199 (139)
  Cycle 1 Day 1, 3 hr n=6,9,4: number analyzed (Participants) | 6 | 9 | 4
  Cycle 1 Day 1, 3 hr n=6,9,4 | 102 (51.8) | 178 (96.3) | 192 (137)
  Cycle 1 Day 1, 4 hr n=6,9,5: number analyzed (Participants) | 6 | 9 | 5
  Cycle 1 Day 1, 4 hr n=6,9,5 | 92.9 (44.0) | 181 (116) | 201 (109)
  Cycle 1 Day 1, 8 hr n=6,9,5: number analyzed (Participants) | 6 | 9 | 5
  Cycle 1 Day 1, 8 hr n=6,9,5 | 75.7 (36.9) | 146 (77.0) | 212 (55.5)
  Cycle 1 Day 2, 24 hr n=6,10,4: number analyzed (Participants) | 6 | 10 | 4
  Cycle 1 Day 2, 24 hr n=6,10,4 | 42.0 (23.7) | 59.7 (49.4) | 95.3 (41.2)
  Cycle 1 Day 5, 0 hr (pre-dose) n=6,7,5: number analyzed (Participants) | 6 | 7 | 5
  Cycle 1 Day 5, 0 hr (pre-dose) n=6,7,5 | 43.5 (42.2) | 88.4 (73.6) | 77.6 (84.2)
  Cycle 1 Day 5,1 hr n=6,6,5: number analyzed (Participants) | 6 | 6 | 5
  Cycle 1 Day 5,1 hr n=6,6,5 | 72.9 (28.3) | 171 (89.8) | 155 (123)
  Cycle 1 Day 5, 2 hr n=6,7,5: number analyzed (Participants) | 6 | 7 | 5
  Cycle 1 Day 5, 2 hr n=6,7,5 | 127 (63.7) | 260 (128) | 324 (112)
  Cycle 1 Day 5, 3 hr n=6,7,5: number analyzed (Participants) | 6 | 7 | 5
  Cycle 1 Day 5, 3 hr n=6,7,5 | 144 (74.6) | 260 (130) | 333 (108)
  Cycle 1 Day 5, 4 hr n=5,7,5: number analyzed (Participants) | 5 | 7 | 5
  Cycle 1 Day 5, 4 hr n=5,7,5 | 133 (67.4) | 226 (111) | 295 (97.9)
  Cycle 1 Day 5, 8 hr n=7,8,3: number analyzed (Participants) | 7 | 8 | 3
  Cycle 1 Day 5, 8 hr n=7,8,3 | 110 (54.3) | 160 (83.1) | 247 (126)
  Cycle 1 Day 6, 24 hr n=7,8,5: number analyzed (Participants) | 7 | 8 | 5
  Cycle 1 Day 6, 24 hr n=7,8,5 | 45.4 (35.9) | 75.1 (66.5) | 72.2 (90.5)
  Cycle 2 Day 1, 0 hr (pre-dose) n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Cycle 2 Day 1, 0 hr (pre-dose) n=4,5,3 | 0 (0) | 0 (0) | 0 (0)
  Cycle 2 Day 1, 1 hr n=5,5,3: number analyzed (Participants) | 5 | 5 | 3
  Cycle 2 Day 1, 1 hr n=5,5,3 | 71.8 (92.9) | 25.5 (28.4) | 32.2 (28.7)
  Cycle 2 Day 1, 2 hr n=5,5,2: number analyzed (Participants) | 5 | 5 | 2
  Cycle 2 Day 1, 2 hr n=5,5,2 | 116 (64.7) | 100 (64.8) | 144 (200)
  Cycle 2 Day 1, 3 hr n=5,5,3: number analyzed (Participants) | 5 | 5 | 3
  Cycle 2 Day 1, 3 hr n=5,5,3 | 111 (58.2) | 146 (99.5) | 178 (147)
  Cycle 2 Day 1, 4 hr n=5,5,3: number analyzed (Participants) | 5 | 5 | 3
  Cycle 2 Day 1, 4 hr n=5,5,3 | 114 (52.8) | 158 (78.4) | 164 (102)
  Cycle 2 Day 1, 8 hr n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Cycle 2 Day 1, 8 hr n=4,5,3 | 90.9 (39.1) | 122 (54.5) | 189 (63.2)
  Cycle 2 Day 2, 24 hr n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Cycle 2 Day 2, 24 hr n=4,5,3 | 67.3 (49.3) | 48.5 (44.2) | 31.7 (5.42)
  Cycle 2 Day 5, 0 hr (pre-dose) n=4,7,3: number analyzed (Participants) | 4 | 7 | 3
  Cycle 2 Day 5, 0 hr (pre-dose) n=4,7,3 | 24.3 (23.8) | 42.5 (50.8) | 29.2 (6.67)
  Cycle 2 Day 5, 3 hr n=3,6,3: number analyzed (Participants) | 3 | 6 | 3
  Cycle 2 Day 5, 3 hr n=3,6,3 | 103 (34.1) | 181 (89.7) | 228 (58.3)
  Cycle 2 Day 6, 24 hr n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Cycle 2 Day 6, 24 hr n=4,5,3 | 34.7 (13.2) | 51.5 (58.3) | 27.5 (6.45)
  Cycle 3 Day 2, 0 hr (pre-dose) n=3,4,4: number analyzed (Participants) | 3 | 4 | 4
  Cycle 3 Day 2, 0 hr (pre-dose) n=3,4,4 | 43.5 (16.5) | 79.1 (96.9) | 39.2 (20.5)
  Cycle 3 Day 5, 0 hr (pre-dose) n=5,6,3: number analyzed (Participants) | 5 | 6 | 3
  Cycle 3 Day 5, 0 hr (pre-dose) n=5,6,3 | 56.8 (47.9) | 81.0 (73.9) | 29.7 (23.3)
  Cycle 4 Day 2, 0 hr (pre-dose) n=5,5,1: number analyzed (Participants) | 5 | 5 | 1
  Cycle 4 Day 2, 0 hr (pre-dose) n=5,5,1 | 36.3 (21.7) | 63.0 (52.4) | 10.9 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 4 Day 5, 0 hr (pre-dose) n=5,6,1: number analyzed (Participants) | 5 | 6 | 1
  Cycle 4 Day 5, 0 hr (pre-dose) n=5,6,1 | 40.4 (29.7) | 50.1 (48.1) | 10.5 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 5 Day 2, 0 hr (pre-dose) n=6,4,4: number analyzed (Participants) | 6 | 4 | 4
  Cycle 5 Day 2, 0 hr (pre-dose) n=6,4,4 | 40.0 (29.3) | 146 (180) | 49.2 (25.1)
  Cycle 5 Day 5, 0 hr (pre-dose) n=6,4,3: number analyzed (Participants) | 6 | 4 | 3
  Cycle 5 Day 5, 0 hr (pre-dose) n=6,4,3 | 78.3 (90.2) | 124 (129) | 32.5 (13.5)
  Cycle 6 Day 2, 0 hr (pre-dose) n=5,2,1: number analyzed (Participants) | 5 | 2 | 1
  Cycle 6 Day 2, 0 hr (pre-dose) n=5,2,1 | 48.0 (28.2) | 60.2 (37.0) | 16.4 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 6 Day 5, 0 hr (pre-dose) n=4,2,1: number analyzed (Participants) | 4 | 2 | 1
  Cycle 6 Day 5, 0 hr (pre-dose) n=4,2,1 | 79.0 (52.2) | 68.9 (68.1) | 9.02 (NA) — Standard deviation was not calculable due to the single data point.

16. Secondary Outcome: Concentration Versus Time Profile for Rineterkib in Part 1
Time Frame: Days 1, 2, 15, and 16 of Cycle 1; Day 1 of Cycles 2, 3, 4, 5, and 6. Each cycle was 28 days.
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ruxolitinib + Rineterkib 200 mg
Number analyzed (Participants) | 9
ng/mL
  Cycle 1 Day 1, 0 hr (pre-dose) n=9 | 0 (0)
  Cycle 1 Day 1, 0.5 hr n=9 | 68.3 (68.8)
  Cycle 1 Day 1, 1 hr n=8: number analyzed (Participants) | 8
  Cycle 1 Day 1, 1 hr n=8 | 235 (343)
  Cycle 1 Day 1, 2 hr n=8: number analyzed (Participants) | 8
  Cycle 1 Day 1, 2 hr n=8 | 340 (229)
  Cycle 1 Day 1, 3 hr n=9 | 352 (244)
  Cycle 1 Day 1, 4 hr n=9 | 325 (173)
  Cycle 1 Day 1, 8 hr n=7: number analyzed (Participants) | 7
  Cycle 1 Day 1, 8 hr n=7 | 244 (128)
  Cycle 1 Day 2, 24 hr n=9 | 261 (419)
  Cycle 1 Day 2, 0 hr (pre-dose) n=8: number analyzed (Participants) | 8
  Cycle 1 Day 2, 0 hr (pre-dose) n=8 | 234 (440)
  Cycle 1 Day 15, 0 hr (pre-dose) n=8: number analyzed (Participants) | 8
  Cycle 1 Day 15, 0 hr (pre-dose) n=8 | 330 (222)
  Cycle 1 Day 15 0.5 hr n=8: number analyzed (Participants) | 8
  Cycle 1 Day 15 0.5 hr n=8 | 581 (464)
  Cycle 1 Day 15, 1 hr n=n=9 | 735 (620)
  Cycle 1 Day 15, 2 hr n=8: number analyzed (Participants) | 8
  Cycle 1 Day 15, 2 hr n=8 | 749 (512)
  Cycle 1 Day 15, 3 hr n=8: number analyzed (Participants) | 8
  Cycle 1 Day 15, 3 hr n=8 | 789 (616)
  Cycle 1 Day 15, 4 hr n=8: number analyzed (Participants) | 8
  Cycle 1 Day 15, 4 hr n=8 | 771 (484)
  Cycle 1 Day 15, 8 hr n=9 | 633 (403)
  Cycle 1 Day 16, 24 hr n=8: number analyzed (Participants) | 8
  Cycle 1 Day 16, 24 hr n=8 | 528 (618)
  Cycle 1 Day 16, 0 hr (pre-dose) n=8: number analyzed (Participants) | 8
  Cycle 1 Day 16, 0 hr (pre-dose) n=8 | 305 (222)
  Cycle 2 Day 1, 0 hr (pre-dose) n=9 | 314 (171)
  Cycle 3 Day 1, 0 hr (pre-dose) n=6: number analyzed (Participants) | 6
  Cycle 3 Day 1, 0 hr (pre-dose) n=6 | 406 (341)
  Cycle 4 Day 1, 0 hr (pre-dose) n=5: number analyzed (Participants) | 5
  Cycle 4 Day 1, 0 hr (pre-dose) n=5 | 402 (364)
  Cycle 5 Day 1, 0 hr (pre-dose) n=3: number analyzed (Participants) | 3
  Cycle 5 Day 1, 0 hr (pre-dose) n=3 | 232 (165)
  Cycle 6 Day 1, 0 hr (pre-dose) n=3: number analyzed (Participants) | 3
  Cycle 6 Day 1, 0 hr (pre-dose) n=3 | 340 (125)

17. Secondary Outcome: Concentration Versus Time Profile for Crizanlizumab in Part 1
Description: EOI = end of infusion
Time Frame: Days 1, 2, 8, and 15 of Cycles 1, 2, and 3; Day 1 of Cycles 4, 5, 6, and 9. Each cycle was 28 days.
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ruxolitinib + Crizanlizumab
Number analyzed (Participants) | 5
ng/mL
  Cycle 1 Day 1, 0 H / PRE-INFUSION n=4: number analyzed (Participants) | 4
  Cycle 1 Day 1, 0 H / PRE-INFUSION n=4 | 0 (0)
  Cycle 1 Day 1, 1H POST EOI n=5 | 114000 (36400)
  Cycle 1 Day 2, 24H POST START OF INFUSION n=4: number analyzed (Participants) | 4
  Cycle 1 Day 2, 24H POST START OF INFUSION n=4 | 78700 (10500)
  Cycle 1 Day 8, 168H POST START OF INFUSION n=5 | 28700 (12200)
  Cycle 1 Day 15, 336H POST START OF INFUSION n=5 | 9280 (4540)
  Cycle 1 Day 15, 0 H / PRE-INFUSION n=1: number analyzed (Participants) | 1
  Cycle 1 Day 15, 0 H / PRE-INFUSION n=1 | 7710 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 2 Day 1, 0 H / PRE-INFUSION n=5 | 20700 (8980)
  Cycle 2 Day 1, 1H POST EOI n=5 | 135000 (43100)
  Cycle 2 Day 1, 336H POST START OF INFUSION n=1,: number analyzed (Participants) | 1
  Cycle 2 Day 1, 336H POST START OF INFUSION n=1, | 15500 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 3 Day 1, 672H POST START OF INFUSION n=5 | 8710 (8350)
  Cycle 3 Day 1, 0 H / PRE-INFUSION n=5 | 8710 (8350)
  Cycle 3 Day 1, 1H POST EOI n=4: number analyzed (Participants) | 4
  Cycle 3 Day 1, 1H POST EOI n=4 | 103000 (59200)
  Cycle 3 Day 2, 24H POST START OF INFUSION n=5 | 95500 (42300)
  Cycle 3 Day 8, 168H POST START OF INFUSION n=5 | 37100 (19400)
  Cycle 3 Day 15, 336H POST START OF INFUSION n=5 | 21000 (17700)
  Cycle 4 Day 1, 672H POST START OF INFUSION n=5 | 5900 (6710)
  Cycle 4 Day 1, 0 H / PRE-INFUSION n=5 | 5900 (6710)
  Cycle 4 Day 1, 1H POST EOI n=5 | 128000 (33200)
  Cycle 5 Day 1, 672H POST START OF INFUSION n=4: number analyzed (Participants) | 4
  Cycle 5 Day 1, 672H POST START OF INFUSION n=4 | 6780 (7830)
  Cycle 5 Day 1, 0 H / PRE-INFUSION n=4: number analyzed (Participants) | 4
  Cycle 5 Day 1, 0 H / PRE-INFUSION n=4 | 6780 (7830)
  Cycle 5 Day 1, 1H POST EOI n=3: number analyzed (Participants) | 3
  Cycle 5 Day 1, 1H POST EOI n=3 | 122000 (29400)
  Cycle 6 Day 1, 672H POST START OF INFUSION n=4: number analyzed (Participants) | 4
  Cycle 6 Day 1, 672H POST START OF INFUSION n=4 | 6930 (8000)
  Cycle 6 Day 1, 0 H / PRE-INFUSION n=4: number analyzed (Participants) | 4
  Cycle 6 Day 1, 0 H / PRE-INFUSION n=4 | 6930 (8000)
  Cycle 6 Day 1, 1H POST EOI n=4: number analyzed (Participants) | 4
  Cycle 6 Day 1, 1H POST EOI n=4 | 128000 (39600)
  Cycle 9 Day 1, 0 H / PRE-INFUSION n=3: number analyzed (Participants) | 3
  Cycle 9 Day 1, 0 H / PRE-INFUSION n=3 | 5500 (9530)

18. Secondary Outcome: Concentration Versus Time Profile for Sabatolimab in Part 1
Description: EOI = end of infusion
Time Frame: Days 1, 2, 8, and 15 of Cycles 1, 2, and 3; Day 1 of Cycles 4 and 5. Each cycle was 28 days.
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ruxolitinib + Sabatolimab
Number analyzed (Participants) | 2
ng/mL
  Cycle 1 Day 1, 0 H / PRE-INFUSION n=2 | 0 (0)
  Cycle 1 Day 1, 1H POST EOI n=1: number analyzed (Participants) | 1
  Cycle 1 Day 1, 1H POST EOI n=1 | 143 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 1 Day 2, 24H POST START OF INFUSION n=2 | 109 (13.2)
  Cycle 1 Day 8, 168H POST START OF INFUSION n=1: number analyzed (Participants) | 1
  Cycle 1 Day 8, 168H POST START OF INFUSION n=1 | 57.0 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 1 Day 15, 336H POST START OF INFUSION n=2 | 41.8 (7.28)
  Cycle 2 Day 1, 672H POST START OF INFUSION n=2 | 16.1 (9.16)
  Cycle 2 Day 1, 0 H / PRE-INFUSION n=2 | 16.1 (9.16)
  Cycle 2 Day 1, 1H POST EOI n=1: number analyzed (Participants) | 1
  Cycle 2 Day 1, 1H POST EOI n=1 | 126 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 3 Day 1, 672H POST START OF INFUSION n=2 | 26.0 (5.09)
  Cycle 3 Day 1, 0 H / PRE-INFUSION n=2 | 26.0 (5.09)
  Cycle 3 Day 1, 1H POST EOI n=2 | 150 (33.2)
  Cycle 3 Day 2, 24H POST START OF INFUSION n=2 | 125 (10.6)
  Cycle 3 Day 8, 168H POST START OF INFUSION n=2 | 80.5 (19.1)
  Cycle 3 Day 15, 336H POST START OF INFUSION n=2 | 58.0 (12.3)
  Cycle 4 Day 1, 672H POST START OF INFUSION n=1: number analyzed (Participants) | 1
  Cycle 4 Day 1, 672H POST START OF INFUSION n=1 | 31.1 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 4 Day 1, 0 H / PRE-INFUSION n=2 | 30.0 (1.56)
  Cycle 4 Day 1, 1H POST EOI n=2 | 141 (11.3)
  Cycle 5 Day 1, 0 H / PRE-INFUSION n=2 | 32.9 (3.82)
  Cycle 5 Day 1, 1H POST EOI n=2 | 152 (9.19)

19. Secondary Outcome: Concentration Versus Time Profile for NIS793 in Part 1
Description: EOI = end of infusion
Time Frame: Days 1, 2, 4, 8, 11, and 15 of Cycles 1, 2, and 3; Day 1 of Cycles 4 and 5. Each cycle was 28 days.
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 4
ng/mL
  Cycle 1 Day 1, 0 H / PRE-INFUSION n=4 | 0 (0)
  Cycle 1 Day 1, 1H POST EOI n=4 | 439000 (56100)
  Cycle 1 Day 2, 24H POST START OF INFUSION n=4 | 349000 (52800)
  Cycle 1 Day 4, 72H POST START OF INFUSION n=4 | 279000 (48400)
  Cycle 1 Day 8, 168H POST START OF INFUSION n=3: number analyzed (Participants) | 3
  Cycle 1 Day 8, 168H POST START OF INFUSION n=3 | 196000 (31000)
  Cycle 1 Day 11, 240H POST START OF INFUSION n=4 | 183000 (45400)
  Cycle 1 Day 15, 336H POST START OF INFUSION n=4 | 161000 (37500)
  Cycle 2 Day 1, 504H POST START OF INFUSION n=4 | 132000 (33300)
  Cycle 2 Day 1, 0 H / PRE-INFUSION n=4 | 132000 (33300)
  Cycle 3 Day 1, 0 H / PRE-INFUSION n=3: number analyzed (Participants) | 3
  Cycle 3 Day 1, 0 H / PRE-INFUSION n=3 | 187000 (61000)
  Cycle 3 Day 1, 1H POST EOI n=3: number analyzed (Participants) | 3
  Cycle 3 Day 1, 1H POST EOI n=3 | 743000 (314000)
  Cycle 3 Day 2, 24H POST START OF INFUSION n=2: number analyzed (Participants) | 2
  Cycle 3 Day 2, 24H POST START OF INFUSION n=2 | 632000 (17000)
  Cycle 3 Day 4, 72H POST START OF INFUSION n=3: number analyzed (Participants) | 3
  Cycle 3 Day 4, 72H POST START OF INFUSION n=3 | 448000 (114000)
  Cycle 3 Day 8, 168H POST START OF INFUSION n=3: number analyzed (Participants) | 3
  Cycle 3 Day 8, 168H POST START OF INFUSION n=3 | 383000 (103000)
  Cycle 3 Day 11, 240H POST START OF INFUSION n=2: number analyzed (Participants) | 2
  Cycle 3 Day 11, 240H POST START OF INFUSION n=2 | 262000 (93300)
  Cycle 3 Day 15, 336H POST START OF INFUSION n=3: number analyzed (Participants) | 3
  Cycle 3 Day 15, 336H POST START OF INFUSION n=3 | 265000 (51500)
  Cycle 4 Day 1, 504H POST START OF INFUSION n=1: number analyzed (Participants) | 1
  Cycle 4 Day 1, 504H POST START OF INFUSION n=1 | 281000 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 4 Day 1, 0 H / PRE-INFUSION n=2: number analyzed (Participants) | 2
  Cycle 4 Day 1, 0 H / PRE-INFUSION n=2 | 232000 (70000)
  Cycle 5 Day 1, 0 H / PRE-INFUSION n=1: number analyzed (Participants) | 1
  Cycle 5 Day 1, 0 H / PRE-INFUSION n=1 | 280000 (NA) — Standard deviation was not calculable due to the single data point.

20. Secondary Outcome: Concentration Versus Time Profile for Ruxolitinib in Part 1
Time Frame: Days 1, 2, 5, 6, and 15 of Cycles 1 and 2; Day 16 of Cycle 1; Days 1, 2, and 15 of Cycle 3; Days 1 and 5 of Cycles 4, 5, and 6. Each cycle was 28 days.
Population: The pharmacokinetic (PK) analysis set included all enrolled subjects who had an evaluable PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793
Number analyzed (Participants) | 7 | 8 | 6 | 8 | 4 | 2 | 4
ng/mL
  Cycle 1 Day 1, 0 hr (pre-dose) n=6,6,5,7,3,2,4: number analyzed (Participants) | 6 | 6 | 5 | 7 | 3 | 2 | 4
  Cycle 1 Day 1, 0 hr (pre-dose) n=6,6,5,7,3,2,4 | 34.7 (17.8) | 21.3 (14.5) | 11.8 (13.4) | 20.1 (16.1) | 12.9 (6.31) | 51.2 (61.0) | 37.9 (48.4)
  Cycle 1 Day 1, 0.5 hr n=6,5,6,8,2,2,3: number analyzed (Participants) | 6 | 5 | 6 | 8 | 2 | 2 | 3
  Cycle 1 Day 1, 0.5 hr n=6,5,6,8,2,2,3 | 284 (128) | 152 (91.1) | 95.7 (63.2) | 185 (100) | 107 (119) | 57.1 (44.0) | 108 (128)
  Cycle 1 Day 1, 1 hr n=6,6,6,7,2,2,3: number analyzed (Participants) | 6 | 6 | 6 | 7 | 2 | 2 | 3
  Cycle 1 Day 1, 1 hr n=6,6,6,7,2,2,3 | 240 (78.9) | 167 (51.7) | 124 (64.5) | 192 (106) | 65.7 (59.9) | 110 (44.1) | 164 (140)
  Cycle 1 Day 1, 2 hr n=6,6,6,7,2,2,3: number analyzed (Participants) | 6 | 6 | 6 | 7 | 2 | 2 | 3
  Cycle 1 Day 1, 2 hr n=6,6,6,7,2,2,3 | 174 (55.3) | 143 (48.6) | 98.9 (46.2) | 140 (112) | 170 (140) | 72.7 (4.10) | 187 (105)
  Cycle 1 Day 1, 3 hr n=6,6,5,8,2,2,3: number analyzed (Participants) | 6 | 6 | 5 | 8 | 2 | 2 | 3
  Cycle 1 Day 1, 3 hr n=6,6,5,8,2,2,3 | 125 (36.6) | 114 (42.1) | 62.4 (31.1) | 97.4 (75.7) | 124 (91.0) | 54.4 (10.4) | 184 (77.9)
  Cycle 1 Day 1, 4 hr n=6,6,6,8,2,2,3: number analyzed (Participants) | 6 | 6 | 6 | 8 | 2 | 2 | 3
  Cycle 1 Day 1, 4 hr n=6,6,6,8,2,2,3 | 93.2 (26.5) | 77.8 (40.0) | 50.2 (23.4) | 59.2 (46.1) | 101 (81.2) | 28.3 (7.28) | 190 (58.4)
  Cycle 1 Day 1, 8 hr n=6,6,6,8,4,2,3: number analyzed (Participants) | 6 | 6 | 6 | 8 | 4 | 2 | 3
  Cycle 1 Day 1, 8 hr n=6,6,6,8,4,2,3 | 51.6 (18.7) | 32.2 (19.1) | 24.0 (15.0) | 29.9 (19.8) | 39.5 (29.2) | 7.75 (1.52) | 44.4 (35.3)
  Cycle 1 Day 2, 0 hr (pre-dose) n=7,6,4,8,1,1,0: number analyzed (Participants) | 7 | 6 | 4 | 8 | 1 | 1 | 0
  Cycle 1 Day 2, 0 hr (pre-dose) n=7,6,4,8,1,1,0 | 18.2 (13.0) | 13.4 (11.1) | 11.2 (16.2) | 17.6 (19.9) | 30.3 (NA) — Standard deviation was not calculable due to the single data point. | 0 (NA) — Standard deviation was not calculable due to the single data point. |
  Cycle 1 Day 5, 0 hr (pre-dose) n=6,8,6,0,0,0,0: number analyzed (Participants) | 6 | 8 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 5, 0 hr (pre-dose) n=6,8,6,0,0,0,0 | 15.5 (13.9) | 14.7 (14.0) | 9.33 (10.6) |  |  |  |
  Cycle 1 Day 5, 1 hr n=6,7,6,0,0,0,0: number analyzed (Participants) | 6 | 7 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 5, 1 hr n=6,7,6,0,0,0,0 | 160 (79.5) | 221 (83.7) | 130 (66.6) |  |  |  |
  Cycle 1 Day 5, 2 hr n=6,8,6,0,0,0,0: number analyzed (Participants) | 6 | 8 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 5, 2 hr n=6,8,6,0,0,0,0 | 149 (64.0) | 140 (45.6) | 90.0 (41.4) |  |  |  |
  Cycle 1 Day 5, 3 hr n=6,8,6,0,0,0,0: number analyzed (Participants) | 6 | 8 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 5, 3 hr n=6,8,6,0,0,0,0 | 104 (45.2) | 100 (39.1) | 61.8 (31.7) |  |  |  |
  Cycle 1 Day 5, 4 hr n=6,8,6,0,0,0,0: number analyzed (Participants) | 6 | 8 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 5, 4 hr n=6,8,6,0,0,0,0 | 81.4 (38.4) | 71.2 (30.1) | 34.1 (16.1) |  |  |  |
  Cycle 1 Day 5, 8 hr n=6,8,4,0,0,0,0: number analyzed (Participants) | 6 | 8 | 4 | 0 | 0 | 0 | 0
  Cycle 1 Day 5, 8 hr n=6,8,4,0,0,0,0 | 37.6 (22.6) | 22.9 (13.7) | 16.2 (13.4) |  |  |  |
  Cycle 1 Day 6, 0 hr (pre-dose) n=6,7,5,0,0,0,0: number analyzed (Participants) | 6 | 7 | 5 | 0 | 0 | 0 | 0
  Cycle 1 Day 6, 0 hr (pre-dose) n=6,7,5,0,0,0,0 | 11.5 (12.1) | 37.8 (63.4) | 6.28 (9.31) |  |  |  |
  Cycle 1 Day 15, 0 hr (pre-dose) n=7,8,4,7,3,2,0: number analyzed (Participants) | 7 | 8 | 4 | 7 | 3 | 2 | 0
  Cycle 1 Day 15, 0 hr (pre-dose) n=7,8,4,7,3,2,0 | 23.2 (34.0) | 23.6 (19.8) | 11.2 (17.4) | 11.9 (14.2) | 12.6 (10.1) | 4.06 (2.28) |
  Cycle 1 Day 15, 0.5 hr n=0,0,0,7,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 7 | 0 | 0 | 0
  Cycle 1 Day 15, 0.5 hr n=0,0,0,7,0,0,0 |  |  |  | 231 (115) |  |  |
  Cycle 1 Day 15, 1 hr n=0,0,0,8,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 8 | 0 | 0 | 0
  Cycle 1 Day 15, 1 hr n=0,0,0,8,0,0,0 |  |  |  | 194 (139) |  |  |
  Cycle 1 Day 15, 2 hr n=0,0,0,7,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 7 | 0 | 0 | 0
  Cycle 1 Day 15, 2 hr n=0,0,0,7,0,0,0 |  |  |  | 126 (58.7) |  |  |
  Cycle 1 Day 15, 3 hr n=0,0,0,7,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 7 | 0 | 0 | 0
  Cycle 1 Day 15, 3 hr n=0,0,0,7,0,0,0 |  |  |  | 103 (59.6) |  |  |
  Cycle 1 Day 15, 4 hr n=0,0,0,7,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 7 | 0 | 0 | 0
  Cycle 1 Day 15, 4 hr n=0,0,0,7,0,0,0 |  |  |  | 76.3 (53.5) |  |  |
  Cycle 1 Day 15, 8 hr n=0,0,0,8,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 8 | 0 | 0 | 0
  Cycle 1 Day 15, 8 hr n=0,0,0,8,0,0,0 |  |  |  | 27.9 (21.7) |  |  |
  Cycle 1 Day 16, 0 hr (pre-dose) n=0,0,0,6,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 6 | 0 | 0 | 0
  Cycle 1 Day 16, 0 hr (pre-dose) n=0,0,0,6,0,0,0 |  |  |  | 14.4 (15.2) |  |  |
  Cycle 2 Day 1, 0 hr (pre-dose) n=6,7,5,8,4,2,3: number analyzed (Participants) | 6 | 7 | 5 | 8 | 4 | 2 | 3
  Cycle 2 Day 1, 0 hr (pre-dose) n=6,7,5,8,4,2,3 | 25.9 (23.4) | 19.3 (18.8) | 11.4 (20.7) | 45.7 (108) | 13.7 (4.84) | 28.4 (39.1) | 65.1 (88.9)
  Cycle 2 Day 1, 1 hr n=6,7,5,0,0,0,0: number analyzed (Participants) | 6 | 7 | 5 | 0 | 0 | 0 | 0
  Cycle 2 Day 1, 1 hr n=6,7,5,0,0,0,0 | 212 (89.8) | 186 (113) | 114 (82.4) |  |  |  |
  Cycle 2 Day 1, 2 hr n=6,7,4,0,0,0,0: number analyzed (Participants) | 6 | 7 | 4 | 0 | 0 | 0 | 0
  Cycle 2 Day 1, 2 hr n=6,7,4,0,0,0,0 | 144 (76.0) | 165 (82.2) | 56.2 (30.9) |  |  |  |
  Cycle 2 Day 1, 3 hr n=6,7,5,0,0,0,0: number analyzed (Participants) | 6 | 7 | 5 | 0 | 0 | 0 | 0
  Cycle 2 Day 1, 3 hr n=6,7,5,0,0,0,0 | 108 (50.8) | 127 (61.7) | 50.3 (26.4) |  |  |  |
  Cycle 2 Day 1, 4 hr n=5,7,5,0,0,0,0: number analyzed (Participants) | 5 | 7 | 5 | 0 | 0 | 0 | 0
  Cycle 2 Day 1, 4 hr n=5,7,5,0,0,0,0 | 89.9 (39.8) | 106 (39.5) | 45.6 (25.8) |  |  |  |
  Cycle 2 Day 1, 8 hr n=4,6,5,0,0,0,0: number analyzed (Participants) | 4 | 6 | 5 | 0 | 0 | 0 | 0
  Cycle 2 Day 1, 8 hr n=4,6,5,0,0,0,0 | 47.3 (31.5) | 45.8 (19.4) | 30.9 (28.1) |  |  |  |
  Cycle 2 Day 2, 0 hr (pre-dose) n=3,6,5,0,0,0,0: number analyzed (Participants) | 3 | 6 | 5 | 0 | 0 | 0 | 0
  Cycle 2 Day 2, 0 hr (pre-dose) n=3,6,5,0,0,0,0 | 74.0 (62.3) | 19.2 (19.7) | 13.9 (20.5) |  |  |  |
  Cycle 2 Day 5, 0 hr (pre-dose) n=3,8,4,0,0,0,0: number analyzed (Participants) | 3 | 8 | 4 | 0 | 0 | 0 | 0
  Cycle 2 Day 5, 0 hr (pre-dose) n=3,8,4,0,0,0,0 | 15.4 (6.29) | 15.2 (11.3) | 4.45 (4.57) |  |  |  |
  Cycle 2 Day 6, 0 hr (pre-dose) n=4,5,4,0,0,0,0: number analyzed (Participants) | 4 | 5 | 4 | 0 | 0 | 0 | 0
  Cycle 2 Day 6, 0 hr (pre-dose) n=4,5,4,0,0,0,0 | 7.36 (7.32) | 46.8 (80.0) | 2.40 (2.74) |  |  |  |
  Cycle 2 Day 15, 0 hr (pre-dose) n=6,8,3,0,1,2,0: number analyzed (Participants) | 6 | 8 | 3 | 0 | 1 | 2 | 0
  Cycle 2 Day 15, 0 hr (pre-dose) n=6,8,3,0,1,2,0 | 22.4 (17.2) | 22.1 (22.7) | 1.93 (1.65) |  | 63.6 (NA) — Standard deviation was not calculable due to the single data point. | 7.95 (8.14) |
  Cycle 3 Day 1, 0 hr (pre-dose) n=7,7,4,6,4,2,2: number analyzed (Participants) | 7 | 7 | 4 | 6 | 4 | 2 | 2
  Cycle 3 Day 1, 0 hr (pre-dose) n=7,7,4,6,4,2,2 | 24.2 (15.5) | 23.2 (21.8) | 4.50 (4.03) | 11.1 (10.9) | 12.0 (6.36) | 2.44 (1.46) | 84.6 (96.8)
  Cycle 3 Day 2, 0 hr (pre-dose) n=5,6,3,0,0,0,0: number analyzed (Participants) | 5 | 6 | 3 | 0 | 0 | 0 | 0
  Cycle 3 Day 2, 0 hr (pre-dose) n=5,6,3,0,0,0,0 | 12.6 (13.9) | 31.9 (38.9) | 2.33 (1.57) |  |  |  |
  Cycle 3 Day 15, 0 hr (pre-dose) n=5,5,2,0,4,2,0: number analyzed (Participants) | 5 | 5 | 2 | 0 | 4 | 2 | 0
  Cycle 3 Day 15, 0 hr (pre-dose) n=5,5,2,0,4,2,0 | 18.7 (18.4) | 45.2 (41.5) | 3.95 (4.10) |  | 10.9 (6.89) | 12.5 (9.14) |
  Cycle 4 Day 1, 0 hr (pre-dose) n=7,5,3,5,4,1,1: number analyzed (Participants) | 7 | 5 | 3 | 5 | 4 | 1 | 1
  Cycle 4 Day 1, 0 hr (pre-dose) n=7,5,3,5,4,1,1 | 17.5 (18.2) | 20.9 (22.2) | 4.53 (6.44) | 18.2 (33.8) | 14.0 (7.81) | 2.94 (NA) — Standard deviation was not calculable due to the single data point. | 24.4 (NA) — Standard deviation was not calculable due to the single data point.
  Cycle 4 Day 5, 0 hr (pre-dose) n=5,6,3,0,0,0,0: number analyzed (Participants) | 5 | 6 | 3 | 0 | 0 | 0 | 0
  Cycle 4 Day 5, 0 hr (pre-dose) n=5,6,3,0,0,0,0 | 13.6 (13.7) | 9.12 (13.5) | 7.99 (11.4) |  |  |  |
  Cycle 5 Day 1, 0 hr (pre-dose) n=7,6,4,3,3,0,0: number analyzed (Participants) | 7 | 6 | 4 | 3 | 3 | 0 | 0
  Cycle 5 Day 1, 0 hr (pre-dose) n=7,6,4,3,3,0,0 | 16.4 (16.1) | 12.7 (12.0) | 5.30 (5.94) | 10.3 (13.6) | 20.1 (23.0) |  |
  Cycle 5 Day 5, 0 hr (pre-dose) n=5,3,3,0,0,0,0: number analyzed (Participants) | 5 | 3 | 3 | 0 | 0 | 0 | 0
  Cycle 5 Day 5, 0 hr (pre-dose) n=5,3,3,0,0,0,0 | 26.6 (16.4) | 9.54 (13.2) | 2.79 (2.46) |  |  |  |
  Cycle 6 Day 1, 0 hr (pre-dose) n=4,4,2,3,3,0,0: number analyzed (Participants) | 4 | 4 | 2 | 3 | 3 | 0 | 0
  Cycle 6 Day 1, 0 hr (pre-dose) n=4,4,2,3,3,0,0 | 15.8 (19.5) | 17.0 (19.7) | 0.608 (0.0672) | 21.9 (23.2) | 27.3 (32.8) |  |
  Cycle 6 Day 5, 0 hr (pre-dose) n=3,4,2,0,0,0,0: number analyzed (Participants) | 3 | 4 | 2 | 0 | 0 | 0 | 0
  Cycle 6 Day 5, 0 hr (pre-dose) n=3,4,2,0,0,0,0 | 24.8 (19.9) | 11.5 (8.34) | 0.957 (0.528) |  |  |  |

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus post-treatment safety follow-up, up to a maximum duration of approximately 44 months.
Groups:
- Part 1: Ruxolitinib + Siremadlin Total: Total
- All Subjects: All Subjects
Arm/Group | Part 1: Ruxolitinib + Siremadlin 20 mg | Part 1: Ruxolitinib + Siremadlin 30 mg | Part 1: Ruxolitinib + Siremadlin 40 mg | Part 1: Ruxolitinib + Siremadlin Total | Part 1: Ruxolitinib + Rineterkib 200 mg | Part 1: Ruxolitinib + Crizanlizumab | Part 1: Ruxolitinib + Sabatolimab | Part 1: Ruxolitinib + NIS793 | Part 2: Ruxolitinib | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10 | 3/6 | 3/23 | 1/9 | 0/6 | 0/2 | 0/4 | 0/1 | 4/45
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/10 | 4/6 | 9/23 | 3/9 | 1/6 | 1/2 | 1/4 | 0/1 | 15/45
Other Adverse Events (participants affected / at risk) | 7/7 | 10/10 | 6/6 | 23/23 | 9/9 | 6/6 | 2/2 | 3/4 | 0/1 | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ruxolitinib + Siremadlin 20 mg (N=7) | Part 1: Ruxolitinib + Siremadlin 30 mg (N=10) | Part 1: Ruxolitinib + Siremadlin 40 mg (N=6) | Part 1: Ruxolitinib + Siremadlin Total (N=23) | Part 1: Ruxolitinib + Rineterkib 200 mg (N=9) | Part 1: Ruxolitinib + Crizanlizumab (N=6) | Part 1: Ruxolitinib + Sabatolimab (N=2) | Part 1: Ruxolitinib + NIS793 (N=4) | Part 2: Ruxolitinib (N=1) | All Subjects (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Product administration error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ruxolitinib + Siremadlin 20 mg (N=7) | Part 1: Ruxolitinib + Siremadlin 30 mg (N=10) | Part 1: Ruxolitinib + Siremadlin 40 mg (N=6) | Part 1: Ruxolitinib + Siremadlin Total (N=23) | Part 1: Ruxolitinib + Rineterkib 200 mg (N=9) | Part 1: Ruxolitinib + Crizanlizumab (N=6) | Part 1: Ruxolitinib + Sabatolimab (N=2) | Part 1: Ruxolitinib + NIS793 (N=4) | Part 2: Ruxolitinib (N=1) | All Subjects (N=45)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 5 | 15 | 1 | 1 | 0 | 2 | 0 | 19
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 8 | 3 | 11 | 0 | 0 | 0 | 0 | 0 | 11
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 7 | 6 | 14 | 2 | 1 | 2 | 0 | 0 | 19
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Presbyopia (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Serous retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 5 | 6 | 2 | 0 | 0 | 0 | 13
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 4 | 3 | 13 | 3 | 2 | 0 | 0 | 0 | 18
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 4
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Discomfort (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 1 | 2 | 8 | 0 | 0 | 0 | 0 | 0 | 8
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 4
Pyrexia (General disorders) | 0 | 3 | 2 | 5 | 1 | 1 | 0 | 1 | 0 | 8
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Amylase increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Blood folate decreased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Blood potassium increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Heart rate decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Heart sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 5
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 5
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 4
Headache (Nervous system disorders) | 3 | 1 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 7
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 1 | 0 | 6
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Trichodysplasia spinulosa (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 5
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04097821/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT04097821/SAP_001.pdf